CLINICAL TRIAL: NCT05029700
Title: The Effect of Trunk Stabilization Training Combined With Aerobic Training on Neuromuscular Parameters and Functional Exercise Capacity in Patients With Multiple Sclerosis
Brief Title: The Effects of Trunk Stabilization and Aerobic Trainings in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02-09
Record Dates: First submitted 2021-07-08; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Physical Therapy
Keywords: balance; strength; endurance; stability; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined exercise group (Experimental): Combined training consists of trunk stabilization training and aerobic training.
  Interventions: Other: Combined exercise training; Other: Aerobic training
- Control group (Active Comparator): Aerobic training was given to the control group.
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Combined exercise training — Combined exercise group (CEG) performed 30 minutes of aerobic training and also received trunk stabilization training in about 30 minutes after a 10-minute resting period. CEG received treatment 2 times a week for 8 weeks. During trunk stabilization training, the participants were taught how to contract the transversus abdominis and multifidus muscles. Due to the progression protocol, endurance levels of trunk muscles were increased by holding each posture for longer periods. The training was started with theraband resistance, which could be repeated between 10-12 repetitions, and the repetition time was increased up to 20. Aerobic training (AT) was given using a treadmill. A heart rate monitor (Polar V800™, Finland) was used by each patient to follow heart rates during the AT. During AT, the target heart rate was calculated as 60-80% of maximum heart rates (MHR). Each exercise session consisted of a 5-minutes warm-up, 20 minutes of walking, and 5 minutes cool down on the treadmill.
  Arms: Combined exercise group
Other: Aerobic training — Control group (CG) performed 30 minutes of aerobic training.CG received treatment 2 times a week for 8 weeks. Aerobic training (AT) was given using a treadmill. A heart rate monitor (Polar V800™, Finland) was used by each patient to follow their heart rates during the AT. During AT, the target heart rate was calculated as 60-80% of maximum heart rates (MHR). Each exercise session consisted of a 5-minutes warm-up, 20 minutes of walking, and 5 minutes cool down on the treadmill.

SUMMARY:
Balance requires many central nervous system controlled functions, and most or all of these functions can be affected by MS, so balance is very often impaired in patients with MS. Core stability is also decreased in patients with MS. Core stability is among the most important factors that ensure the balance and walking of the participants in different environments and conditions during functional activities. In addition to core muscle activity, lower extremity muscle strength and endurance decrease due to the influence of central nervous system and decrease in physical activity. Functional exercise capacity also decreases due to the influence of the central nervous system and the decrease in physical activity in patients with MS.

Despite all these symptoms and the benefits of exercise training, unfortunately, most MS patients are physically inactive, which can initiate a cycle of deconditioning and worsening of symptoms. In the literature, the combined effects of aerobic training and resistance training have been examined, and it has been stated that combining these two trainings will increase the effectiveness on symptoms. In recent years, trunk stabilization training has started to be included in physiotherapy and rehabilitation programs as an alternative method in patients with MS, based on the knowledge that core stability is effective on many functions and symptoms, as well as aerobic and resistance training. Considering that combined training practices are more effective in reducing symptoms, the investigators think that aerobic training and trunk stabilization training may be more effective in reducing symptoms in patients with MS when applied in combination. In addition, when all these studies were examined, the subtypes of MS patients included in the studies were generally not specified. The effects of these trainings on balance, core stability lower extremity muscle strength and endurance, and functional exercise capacity have not been demonstrated in patients with relapsing remitting MS (RR-MS), the most common type of MS disease. Therefore, the aim of this study is to examine the effects of trunk stabilization training combined with aerobic training on balance, core stability, lower extremity muscle strength and endurance, and functional exercise capacity in patients with RR-MS.

DETAILED DESCRIPTION:
This study was carried out with the purpose of examining the effects of trunk stabilization training combined with aerobic training on balance, core stability, lower extremity muscle strength and endurance, and functional exercise capacity in patients with RR-MS.

A total of 20 patients, 10 in each group, were included in the study. Both the combined exercise group and the control group performed 30 minutes of aerobic training. The combined exercise group also received trunk stabilization training after a 10-minute resting period. Both groups received treatment 2 times a week for 8 weeks (in total 16 sessions). The static and dynamic balance were measured using the posturography (Biodex Balance System SDTM) with Postural Stability Test and Limits of Stability Test. Core stability was assessed by core endurance tests using the McGill protocol. Core endurance tests used are flexion endurance test, extension endurance test, and right and left lateral bridge tests. The lower extremity muscle strength and endurance of the patients were determined by evaluating the strength and endurance of the knee flexor and extensor muscles at angular velocities of 60º/sec and 180º/sec. Evaluations were made using the Biodex System 4 (Biodex Corp, Shirley, NY, USA) isokinetic dynamometer. Functional exercise capacity was assessed using the 6-Minute Walking Test (6-MWT) according to criteria set by the American Thoracic Society.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with relapsing-remitting multiple sclerosis disease by a specialist physician
* Not having an MS attack in the last 3 months
* Having a disability level between 1 and 5 according to the Expanded Disability Status Scale
* Not being included in the physiotherapy and rehabilitation program in the last 3 months

Exclusion Criteria:

* Using corticosteroids in the past 4 weeks
* Being pregnant
* Spinal deformities, spinal disc herniation or other spinal pathologies, orthopedic problems related to hip, knee, ankle

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Static balance | 4 weeks
  Static balance was evaluated by Biodex Balance System SD™ (Biodex Medical Systems, Shirley, New York, USA). Postural Stability Test (PST) was used for static balance assessment of the participants.
  PST is assessed, while participants stand on both feet on the firm surface and with eyes open. In the start position, a dot is defined as a symbolic presentation of participants' center of feet pressure positioned in the center of the coordinate axes on the monitor screen. The participants targets on holding the dot at the center. PST provides overall postural stability index score. Lower scores indicated better performance.
Static balance | 4 weeks
  Static balance was evaluated by Biodex Balance System SD™ (Biodex Medical Systems, Shirley, New York, USA). Postural Stability Test (PST) was used for static balance assessment of the participants.
  PST is assessed, while participants stand on both feet on the firm surface and with eyes open. In the start position, a dot is defined as a symbolic presentation of participants' center of feet pressure positioned in the center of the coordinate axes on the monitor screen. The participants targets on holding the dot at the center. PST provides anterior-posterior postural stability index score. Lower scores indicated better performance.
Static balance | 4 weeks
  Static balance was evaluated by Biodex Balance System SD™ (Biodex Medical Systems, Shirley, New York, USA). Postural Stability Test (PST) was used for static balance assessment of the participants.
  PST is assessed, while participants stand on both feet on the firm surface and with eyes open. In the start position, a dot is defined as a symbolic presentation of participants' center of feet pressure positioned in the center of the coordinate axes on the monitor screen. The participants targets on holding the dot at the center. PST provides medial-lateral postural stability index scores. Lower scores indicated better performance.
Dynamic balance | 4 weeks
  Dynamic balance was evaluated by Biodex Balance System SD™ (Biodex Medical Systems, Shirley, New York, USA). Limits of Stability (LOS) Test was used for dynamic balance assessment of the participants.
  LOS Test consists of standing on the platform and leaning in eight directions to make a cursor displayed on the system's screen hit a target. LOS Test provides overall direction control score. Higher scores indicated better performance

SECONDARY OUTCOMES:
Lower extremity muscle strength | 4 weeks
  The lower extremity muscle strength of the participants were determined by evaluating the strength of the knee flexor and extensor muscles at angular velocities of 60º/second and 180º/second. Evaluations were made using the Biodex System 4 (Biodex Corp, Shirley, NY, USA) isokinetic instrument. The tests were repeated on both the dominant and nondominant sides. As a result of the evaluations, peak torque value was obtained at angular velocities of 60º/second and 180º/second.
Lower extremity muscle strength | 4 weeks
  The lower extremity muscle strength of the participants were determined by evaluating the strength of the knee flexor and extensor muscles at angular velocities of 60º/second and 180º/second. Evaluations were made using the Biodex System 4 (Biodex Corp, Shirley, NY, USA) isokinetic instrument. The tests were repeated on both the dominant and nondominant sides. As a result of the evaluations, peak torque/body weight value was obtained at angular velocities of 60º/second and 180º/second.
Lower extremity muscle endurance | 4 weeks
  The lower extremity muscle endurance of the participants were determined by evaluating the endurance of the knee flexor and extensor muscles at angular velocities of 60º/second and 180º/second. Evaluations were made using the Biodex System 4 (Biodex Corp, Shirley, NY, USA) isokinetic instrument. The tests were repeated on both the dominant and nondominant sides. As a result of the evaluations, peak torque value was obtained at angular velocities of 60º/second and 180º/second.
Lower extremity muscle endurance | 4 weeks
  The lower extremity muscle endurance of the participants were determined by evaluating the endurance of the knee flexor and extensor muscles at angular velocities of 60º/second and 180º/second. Evaluations were made using the Biodex System 4 (Biodex Corp, Shirley, NY, USA) isokinetic instrument. The tests were repeated on both the dominant and nondominant sides. As a result of the evaluations, peak torque/body weight value was obtained at angular velocities of 60º/second and 180º/second.

OTHER OUTCOMES:
Core stability | 4 weeks
  Core stability was assessed by core endurance tests using the McGill protocol. Core endurance tests used are flexion endurance test, extension endurance test, and right and left lateral bridge tests. Results were recorded in seconds. The tests were terminated when the test position was disturbed or the participants said they could not continue the test.
The flexor endurance test | 4 weeks
  The participants were positioned. The trunk was at 60º flexion, knees and hips were at 90º flexion position, the arms were bended across the chest with the hands placed on the opposite shoulder, and the feet were fixed. The trunk support was removed, and the participants were asked to maintain their positions for as long as possible. The test was terminated when the participants were no longer able to hold the position.
The extensor endurance test | 4 weeks
  The participants were positioned in the prone position with the pelvis, hip and knees fixed on the treatment table. The trunk and upper extremities were supported by a chair at the same height as the treatment table. The chair was removed, and the participants maintained the horizontal body position for as long as possible with arms crossed over back of the neck. The test was discontinued when the participant fell below the horizontal position.
The side bridge test | 4 weeks
  The participants were positioned in the side-lying position to make the lower arm in vertical position on the ground, the elbow at 90º flexion position, the forearm on treatment table, the top arm bended across the chest with the hand placed on the opposite shoulder, lower extremities in extension, and the top foot in front of the lower foot on the treatment table. The test was stopped when the side-lying position was lost, or when the hips returned to the mat. The test was evaluated both on the right and left sides.
Functional exercise capacity | 4 weeks
  Functional exercise capacity was assessed using the 6-Minute Walking Test according to criteria set by the American Thoracic Society. The participants were asked to walk for six minutes on a straight, uninterrupted 30-meter corridor at the highest speed they felt safe. The participants were informed that the test could be terminated if the participants could not continue the test. Before starting the test, participants' blood pressure, heart rate and fatigue level were evaluated. At the end of the test, blood pressure, heart rate and fatigue level were re-evaluated. At the end of the test, the end point was marked and the walking distance was recorded in meters.
Heart rate | 4 weeks
  Heart rate was evaluated with a polar heart rate monitor (Polar V800™, Kempele, Finland).
Modified Borg scale | 4 weeks
  Fatigue level was evaluated with the Modified Borg scale. The modified Borg scale is a category scale that evaluates fatigue from 0 to 10. Patients were asked to mark the appropriate value for their condition on the scale. Higher test score indicates increased fatigue.
Blood pressure | 4 weeks
  Systolic and diastolic blood pressures were evaluated with a manual sphygmomanometer (Erka Perfect Aneroid, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Taskin Ozkan, doctorate, Principal Investigator — Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation Etlik, Ankara, Turkey, 06010, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided